CLINICAL TRIAL: NCT02019394
Title: Interventional, Open-label Study Investigating the Absolute Bioavailability of Lu AE58054 After Multiple Oral Dosing and a Single Radio-labelled Intravenous Micro-dose as Well as the Contribution of Cytochrome P450 2D6 to the Exposure of Lu AE58054 in Healthy Subjects
Brief Title: Absolute Bioavailability of Lu AE58054 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 14915A; 2012-005646-37 (EudraCT Number)
Record Dates: First submitted 2013-12-18; First posted 2013-12-24 (Estimated); Last update posted 2014-03-21 (Estimated); Status verified 2014-03

CONDITIONS: Healthy
MeSH Terms: interventions — (2-(6-fluoro-1H-indol-3-yl)-ethyl)-(3-(2,2,3,3-tetrafluoropropoxy)benzyl)amine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lu AE58054 (Experimental)
  Interventions: Drug: Lu AE58054

INTERVENTIONS:
Drug: Lu AE58054 — Oral dosing: 90 mg Lu AE58054 as a single dose once and after a 3 days washout period, once daily for 7 days.
  Intravenous dosing: 90 μg/not more than (NMT) 1000 nCi/37 kBq 14C-Lu AE58054 for intravenous infusion once on Day 10.

SUMMARY:
To determine the absolute bioavailability of the Lu AE58054 tablet formulation at steady state

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women aged between 21-55 years (inclusive) and with an BMI in the range 18.5 to 32 kg/m2 (minimum weight 60 kg for men and 55 kg for women).
* The subjects CYP2D6 genotype must be determined before inclusion into the study.
* Women must not be pregnant or lactating.

Exclusion Criteria:

* The subject is, in the opinion of the investigator, unlikely to comply with the protocol or is unsuitable for any reason.

Other inclusion and exclusion criteria may apply.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2013-12; Primary Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Absolute bioavailability: (AUC0-24) Dose oral/(AUC0-inf) Dose IV | Day 10
  Intravenous (IV)
Ratio of (AUC0-24(PM)/AUC0-24(EM)) | Day 10
  Poor Metaboliser (PM); Extensive Metaboliser (EM)

SECONDARY OUTCOMES:
Number and frequency of adverse events | Up to Day 16
  Standard clinical safety assessments
Number of subjects with adverse events | Up to Day 16
  Adverse event monitoring
Risk of Suicidality | Up to Day 16
  Columbia Suicide Severity Rating Scale (C-SSRS) categorisation based on Columbia Classification Algorithm of Suicide Assessment (C-CASA) definitions

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (1):
- GB803, Nottingham, United Kingdom